CLINICAL TRIAL: NCT04629404
Title: A Randomized, Double-Blind, Placebo-Controlled Clinical Trial to Evaluate the Pharmacodynamics/Pharmacokinetics and Safety of Multiple Intramuscular Doses of LY03003 in Patients With Early Parkinson's Disease
Brief Title: A Clinical Trial to Evaluate the Pharmacodynamics/Pharmacokinetics and Safety of LY03003 in Early PD Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Luye Pharma Group Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LY03003/CT-CHN-105
Record Dates: First submitted 2020-11-05; First posted 2020-11-16 (Actual); Last update posted 2020-11-16 (Actual); Status verified 2020-11

CONDITIONS: Parkinson Disease
Keywords: parkinson disease; LY03003
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LY03003 (Experimental)
  Interventions: Drug: LY03003
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: LY03003 — Firstly, intramuscularly inject 14 mg of the study drug once, continue intramuscularly inject 28 mg of the study drug once after being observed for 1 week to confirm safety, continue intramuscularly inject 42 mg of the study drug once after being observed for 1 week to confirm safety, and prepare to enter the maintenance period of 56 mg dose after being observed for 1 week to confirm safety. During the dose maintenance period, 56 mg of the test drug was intramuscularly injected once a week for a total of 4 consecutive doses.
  Arms: LY03003
Drug: Placebo — Firstly, intramuscularly inject 14 mg of the study drug once, continue intramuscularly inject 28 mg of the study drug once after being observed for 1 week to confirm safety, continue intramuscularly inject 42 mg of the study drug once after being observed for 1 week to confirm safety, and prepare to enter the maintenance period of 56 mg dose after being observed for 1 week to confirm safety. During the dose maintenance period, 56 mg of the test drug was intramuscularly injected once a week for a total of 4 consecutive doses.
  Arms: Placebo

SUMMARY:
A Clinical Trial to Evaluate the Pharmacodynamics/Pharmacokinetics and Safety of LY03003 in Early PD Patients

ELIGIBILITY:
Inclusion Criteria:

1. the subject or his legal representative understands and is willing to participate in this clinical study and voluntarily signs and dates the informed consent form;
2. in the judgment of the investigator, the subject or his legal representative is considered trustworthy and able to comply with the study protocol, visit plan or receive the study drug as required;
3. Subjects aged ≥ 30 years at screening (Visit 1), male or female;
4. Meet the UK Brain Bank diagnostic criteria for essential Parkinson's disease, duration of illness ≤ 5 years, the diagnosis is based on the main sign - bradykinesia, plus at least one of the following symptoms: resting tremor, rigidity or postural reflex disorders, and no other known or suspected cause of Parkinson's disease;
5. Hoehn-Yahr stage ≤ 3 (excluding stage 0) in the "on" state;
6. Mini-Mental State Examination (MMSE) ≥ 25 points;
7. At baseline (Visit 2), the Unified Parkinson's Disease Rating Scale (UPDRS) motor score (Part III) in the "on" state is ≥ 10;
8. if the subject is receiving anticholinergic drugs (e.g., methenamine, diphenhydramine, diethylpromethazine, procyclidine, and biperiden), monoamine oxidase B (MAO-B) inhibitors (e.g., selegiline, rasagiline), N-methyl-d-aspartate (NMDA) antagonists (e.g., amantadine), the dose must be stable for at least 28 days before baseline (Visit 2), and the dose must be maintained during the study;
9. Women of childbearing age (do not meet any of the following conditions: cessation of menstruation for ≥ 12 months; or underwent hysterectomy or oophorectomy; or have medically confirmed ovarian failure) or male subjects agree to take reliable contraception (oral contraceptives, use of condoms, abstinence, etc.) throughout the study (screening visit to the end of the study), and screening (Visit 1) and baseline (Visit 2), women of childbearing age pregnancy test results are negative.

Exclusion Criteria:

1. history of pallidotomy, thalamic lesioning, deep brain stimulation or fetal tissue transplantation;
2. suffering from dementia, active mental illness or hallucinations, major depression;
3. Patients receiving dopamine agonist therapy within 28 days before baseline (Visit 2);
4. received levodopa preparations (containing levodopa compound preparations) within 28 days before baseline (Visit 2);
5. received any of the following drugs within 28 days before baseline (Visit 2): amphetamine, metoclopramide, α-methyldopa, anti-schizophrenia drugs, monoamine oxidase A (MAO-A) inhibitors, reserpine, methylphenidate, cloth;
6. Receiving central nervous system active drug treatment (such as sedative hypnotics, antidepressants, anxiolytics), but excluding the baseline (Visit 2) has remained stable for at least 28 days, and may remain stable during the study;
7. Atypical Parkinson's disease symptoms caused by taking drugs (such as metoclopramide, flunarizine), nervous system inherited metabolic diseases (such as Wilson's disease), encephalitis, cerebrovascular disease or degenerative diseases (such as progressive supranuclear palsy);
8. History of epilepsy, or stroke or transient ischemic attack within 1 year before screening (Visit 1);
9. intolerant or allergic to the following antiemetics, such as domperidone, trimethobenzamide, ondansetron, tropisetron, granisetron and gronium;
10. Clinically significant liver dysfunction, defined as total bilirubin > 1.5 times the upper limit of the reference range or alanine aminotransferase (ALT) or aspartate aminotransferase (AST) > 2 times the upper limit of the reference range;
11. Clinically significant renal dysfunction (serum creatinine > 2.0 mg/dL [> 177 μmol/L]);
12. uncontrolled or significant cardiovascular disease, including New York Heart Association (NYHA) class II or higher congestive heart failure, unstable angina, myocardial infarction within 6 months before baseline (Visit 2), or arrhythmia requiring treatment at screening (Visit 1);
13. At screening (Visit 1) and baseline (Visit 2), QTc interval: male > 470 ms, female > 480 ms;
14. History of symptomatic orthostatic hypotension; or a systolic blood pressure decrease of ≥ 20 mmHg or a diastolic blood pressure decrease of ≥ 10 mmHg at 1 or 3 minutes from a recumbent to an upright position at screening (Visit 1) and baseline (Visit 2); or a supine systolic blood pressure < 105 mmHg at screening (Visit 1) and baseline (Visit 2);
15. History of suicide attempt (including actual attempts, interrupted attempts, or failed attempts) or suicidal ideation in the past 6 months, defined as "yes" to question 4 or 5 on the Columbia-Suicide Severity Rating Scale (C-SSRS) at screening (Visit 1);
16. History of narcolepsy;
17. History of alcoholism, drug abuse, or drug abuse within 5 years before screening (Visit 1), defined as alcohol consumption of more than 14 units of alcohol per week (1 unit = 360 ml of beer or 45 ml of spirits with an alcohol content of 40% or 150 ml of wine);
18. Patients with malignant tumors within 5 years before screening (Visit 1), except for adequately treated cervical carcinoma in situ, basal cell or squamous cell carcinoma of the skin, local prostate cancer after radical surgery, and intraductal carcinoma in situ after radical surgery;
19. Pregnant or lactating women;
20. Previous participation in the rotigotine test can not tolerate or poor efficacy; Allergic constitution or known allergy to rotigotine or rotigotine microsphere preparation components;
21. Allergic constitution or known allergy to rotigotine or rotigotine microsphere preparation components;
22. Participated in other drug clinical trials within 3 months before screening (Visit 1);
23. have other clinically significant medical conditions, psychiatric conditions or laboratory abnormalities that may interfere with the ability of the subject to participate in this study as judged by the investigator.

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2018-11-05 (Actual); Primary Completion 2019-03-14 (Actual); Study Completion 2019-03-14 (Actual)

PRIMARY OUTCOMES:
Pharmacodynamic Measures | From titration to dose-maintenance at day 50
  Change from baseline in (II + III) total score, Part II, Part III scores of the UPDRS
Safety Measures | From titration to dose-maintenance at day 50
  Blood Pressure

SECONDARY OUTCOMES:
Cmax,ss | From titration to dose-maintenance at day 50
  Peak concentration

CONTACTS AND LOCATIONS:
Locations (1):
- Shengjing Hospital of China Medical University, Shenyang, China